CLINICAL TRIAL: NCT01229683
Title: Effects of Interscalene Brachial Plexus Nerve Blocks on the Hand and Forearm
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Other Study IDs: Madison Block
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Shoulder Surgery; Interscalene Nerve Block
Keywords: UCSD; Perineural Nerve Block; Shoulder Surgery; Pain; Grip Strength; Sensation; Interscalene Nerve Block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shoulder Surgery: Patients will be given an interscalene nerve block and then strength and sensation of the hand and forearm will be tested to determine if the block is helping to anesthetize these areas.
  Interventions: Procedure: Interscalene Nerve Block

INTERVENTIONS:
Procedure: Interscalene Nerve Block — Patients undergoing shoulder surgery will be given an Interscalene Nerve Block. The patients' strength and sensation in their hand and forearm will be tested to determine if the nerve block is affectively delivering anesthetic to the nerves that serve these areas.

SUMMARY:
Research study to determine the proportion of cases in which an interscalene brachial plexus nerve block produces hand and forearm anesthesia.

DETAILED DESCRIPTION:
This is a research study to prospectively determine the proportion of cases in which an interscalene brachial plexus nerve block produces hand and forearm anesthesia. The investigators will investigate this issue in patients having shoulder and not hand/forearm surgery. We will test hand grip strength and sensation to determine if the hand and forearm are responding to the anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* unilateral orthopedic shoulder surgery
* already desiring an interscalene brachial plexus nerve block for postoperative analgesia with the anesthetic plan including a preoperative interscalene nerve block with mepivacaine

Exclusion Criteria:

* any known contraindication to study medications or testing hand grip strength pre/post-op
* insulin-dependent diabetes mellitus
* neuropathy of any etiology in the affected extremity
* any anticipated incision site apart from the shoulder
* Obesity
* Pregnancy
* Incarceration
* inability to communicate with the investigators and hospital staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist only of patients undergoing orthopedic shoulder surgery.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Centers (Hillcrest and Thornton), San Diego, California, United States